CLINICAL TRIAL: NCT00733226
Title: Phase IV Study of Effect of OM-85 BV (Broncho-Vaxom) on Wheezing Related Morbidity in Children With Recurrent Wheezing
Brief Title: Effect of OM-85 BV on Wheezing Related Morbidity in Children With Recurrent Wheezing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kecioren Education and Training Hospital (Other)
Responsible Party: Principal Investigator, Cem Hasan Razi, MD, Kecioren Education and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: B100İEG0110001 - 2860
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Results first posted 2010-08-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Asthma
Keywords: wheezing; asthma; childhood; OM-85 BV; Broncho-Vaxom
MeSH Terms: conditions — Asthma; Respiratory Sounds | interventions — Broncho-Vaxom

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Broncho-Vaxom (Active Comparator): The children received one capsule per oral, OM-85 BV (3.5 mg) per day for the first 10 consecutive days of each month for 3 consecutive months.
  Interventions: Drug: OM-85 BV (Broncho-Vaxom)
- 2 (Placebo OM-85 BV) (Placebo Comparator): The children received one capsule per oral, placebo per day for the first 10 consecutive days of each month for 3 consecutive months.
  Interventions: Drug: OM-85 BV (placebo)

INTERVENTIONS:
Drug: OM-85 BV (Broncho-Vaxom) — 3.5 mg capsule, 1 capsule per day for first 10 day of the month, for 3 months
  Other Names: Bronchovaxom 3.5 mg capsule
  Arms: 1 Broncho-Vaxom
Drug: OM-85 BV (placebo) — 3.5 mg oral placebo capsule, 1 placebo capsule per day for first 10 days of the months for 3 months
  Other Names: Bronchovaxom 3.5 mg placebo capsule
  Arms: 2 (Placebo OM-85 BV)

SUMMARY:
The purpose of this study is to determine whether OM-85 BV (Broncho-Vaxom)has any effect on respiratory infections, infection related wheezing attacks, beta-2 agonist use, duration of attacks and effect on serum cytokine levels.

DETAILED DESCRIPTION:
Context: Respiratory infections are the major cause of wheezing attacks in children with recurrent wheezing or asthma in preschool age. OM-85 BV is an bacteria lysate which has been proven to prevent respiratory infections about 40 percent in children.

Objective: To determine if using OM-85 BV diminish the number and duration of the respiratory infections and respiratory infection related wheezing attacks,beta-2 agonist and steroid use, and number and duration of hospitalizations in children with recurrent wheezing and asthma. And also to determine if OM-85 BV has any effect on serum cytokine levels after 6 months.

Study Design/Setting/Participants: A double-blind, randomized, controlled trial of OM-85 BV versus placebo for children 6 months to 6 years of age who have respiratory tract infection related recurrent wheezing attacks.

Intervention: Participants will receive either active Broncho-Vaxom or placebo for 3 months.

Study Measures: They follow up for 1 year for number and duration of wheezing attacks, number, type and duration of respiratory infections, number and duration of beta-2 agonist use, number and duration of steroid use and number and duration of hospitalizations. Serum cytokine levels will measure to determine if Broncho-Vaxom has any effect on serum cytokine levels (at the beginning of the trial and sixth months of the trial).

ELIGIBILITY:
Inclusion Criteria:

* Children with recurrent wheezing who had at least 3 wheezing attacks in the last 6 months
* Children with asthma who had at least 3 wheezing attacks in the last 6 months

Exclusion Criteria:

* Chronic lung disease
* Immun deficiency
* Malabsorption
* Anatomic abnormalities of the respiratory tract
* Gastroesophageal reflux disease

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2007-08; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C H RAZI, MD, Study Director — Kecioren Education and Training Hospital; C H Razi, MD, Principal Investigator — Kecioren Education and Training Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Kecioren Education and Training Hospital, Ankara, Kec.oren
  - Keçiören Education and Training Hospital, Ankara, Keçiören

REFERENCES:
- [Background] Razi CH, Harmanci K, Abaci A, Ozdemir O, Hizli S, Renda R, Keskin F. The immunostimulant OM-85 BV prevents wheezing attacks in preschool children. J Allergy Clin Immunol. 2010 Oct;126(4):763-9. doi: 10.1016/j.jaci.2010.07.038. PMID 20920766

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a randomized, double-blind, placebo-controlled, parallel group study with OM-85 (Broncho-Vaxom; OM PHARMA; Meyrin/Geneva, Switzerland) in patients with recurrent wheezing and performed between August 2007- September 2008 in the outpatient department of Pediatric Allergy of Kecioren Education and Research Hospital in Ankara, Turkey.
Pre-assignment Details: This study comprise 3 months of active treatment and 9 months of follow-up. Duration of the trial was 12 months.
  Eighty of 100 children were selected to enter the trial. 20 children were not included in to the study because of not meeting the inclusion criteria.
Groups:
- Broncho-Vaxom Group: The children received one capsule per oral, OM-85 BV (3.5 mg) per day for the first 10 consecutive days of each month for 3 consecutive months.
- Placebo Group: The children received one capsule per oral, placebo per day for the first 10 consecutive days of each month for 3 consecutive months.
Period: Overall Study
Arm/Group | Broncho-Vaxom Group | Placebo Group
Started | 40 | 40
Completed | 35 | 40
Not Completed | 5 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — moved to another place | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Broncho-Vaxom Group: This group consists of 35 children with recurrent wheezing who received one capsule per oral, OM-85 BV (3.5 mg) per day for the first 10 consecutive days of each month for 3 consecutive months.
- Placebo Group: This group consists of 40 children with recurrent wheezing who received one capsule per oral, placebo per day for the first 10 consecutive days of each month for 3 consecutive months.
- Total: Total of all reporting groups
Arm/Group | Broncho-Vaxom Group | Placebo Group | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 40 | 40 | 80
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.51 (1.48) | 2.65 (1.69) | 2.59 (0.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 28 | 27 | 55
Region of Enrollment [Number; unit: participants]
  Turkey | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Mean Rate of Wheezing Attacks
Description: Acute wheezing attack was defined as episode of progressive increase in shortness of breath, cough, wheezing, retraction of the chest and chest tightness, or combination of these symptoms. When wheezing attack occured it was Over the 12 months of the study mean number (rate) of wheezing attacks/per patient was calculated and compared with placebo. This outcome measure was calculated by dividing cumulative wheezing attacks to number of participants in each group.
Time Frame: 12 months
Measure: Mean (Standard Error); unit: wheezing attacks/per patient
Arm/Group | Broncho-Vaxom Group | Placebo Group
Number analyzed (Participants) | 35 | 40
wheezing attacks/per patient | 3.57 (1.61) | 5.72 (2.72)
Statistical Analysis 1: Comparison: Broncho-Vaxom Group vs Placebo Group; The sample size was computed to prove that a 30% decrease of the rate of virus provoked wheezing attacks in the OM-85 group compared with placebo is statistically significant. Approximately 29 analyzable participants in each group were required, with α=0.05 and β=0.10 (ie, with a power of 90%), respectively. The difference of 30% was taken from both pilot study and clinical experience. Sample size estimation was performed by using NCSS and PASS 2000 software; Test type: Superiority or Other; p = 0.05, Wilcoxon (Mann-Whitney) — P value was not need to adjusted for multiple comparisons; Mean Difference (Final Values) = -2.15, 95% CI 2-sided [-3.20 to -1.10], Standard Error of Mean 0.52

2. Secondary Outcome: Mean Duration (in Day) of Wheezing Attacks Per Patient
Description: Over the 12 months of the study we calculated mean duration of each wheezing attacks/per patients.This measure was calculated separately for each participants by dividing duration of wheezing attacks to number of wheezing attacks.
Time Frame: 12 months
Measure: Mean (Standard Error); unit: day/per patient
Arm/Group | Broncho-Vaxom Group | Placebo Group
Number analyzed (Participants) | 35 | 40
day/per patient | 5.57 (0.35) | 7.66 (0.33)
Statistical Analysis 1: Comparison: Broncho-Vaxom Group vs Placebo Group; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P value was not need to adjusted for multiple comparisons; Mean Difference (Final Values) = -2.08, 95% CI 2-sided [-3.06 to -1.01], Standard Error of Mean 0.49

3. Secondary Outcome: Number of Common Cold
Description: All the common colds were recorded during the 12 months of the study. At the and of the study period the two groups were compared according to the number of common-cold/per patient over the 12 months of the trial.
  This outcome was calculated by dividing cumulative number of common colds by number of participants in each group over the 12 months of the trial.
Time Frame: 12 months
Measure: Mean (Standard Error); unit: common cold/per patients
Arm/Group | Broncho-Vaxom Group | Placebo Group
Number analyzed (Participants) | 35 | 40
common cold/per patients | 3.51 (0.26) | 5.62 (0.31)
Statistical Analysis 1: Comparison: Broncho-Vaxom Group vs Placebo Group; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); P value was not need to adjusted for multiple comparisons; Median Difference (Final Values) = -2.11, 95% CI 2-sided [-2.94 to -1.27], Standard Error of Mean 0.41

4. Secondary Outcome: Number of Wheezing Attacks That Required Systemic Steroid Therapy
Description: All the wheezing attacks which were enough severe to require systemic steroid therapy were recorded over the 12 months of the study.
  At the and of the study period, number of wheezing attacks that required systemic steroid therapy/per patients were calculated. This outcome was calculated by dividing cumulative number of wheezing attacks that required systemic steroid therapy by number of participants in each group.
Time Frame: 12 months
Measure: Mean (Standard Error); unit: wheezing attacks/per patient
Arm/Group | Broncho-Vaxom Group | Placebo Group
Number analyzed (Participants) | 35 | 40
wheezing attacks/per patient | 0.57 (0.14) | 0.90 (0.16)
Statistical Analysis 1: Comparison: Broncho-Vaxom Group vs Placebo Group; Test type: Superiority or Other; p = 0.110, Wilcoxon (Mann-Whitney) — P value was not need to adjusted for multiple comparisons; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-0.77 to 0.11], Standard Error of Mean 0.22

5. Secondary Outcome: Number of Hospitalizations
Description: During the study period of 12 months all hospitalizations for wheezing attacks were recorded.
  Over the 12 months of the trial mean number of hospitalizations/per patients were calculated.
  This outcome was calculated by dividing cumulative number of hospitalizations by number of participants in each group over the 12 months of the trial.
Time Frame: 12 months
Measure: Mean (Standard Error); unit: hospitalization/per patient
Arm/Group | Broncho-Vaxom Group | Placebo Group
Number analyzed (Participants) | 35 | 40
hospitalization/per patient | 0.14 (0.05) | 0.40 (0.12)
Statistical Analysis 1: Comparison: Broncho-Vaxom Group vs Placebo Group; Test type: Superiority or Other; p = 0.195, Wilcoxon (Mann-Whitney) — P value was not need to adjusted for multiple comparisons; Median Difference (Final Values) = -0.25, 95% CI 2-sided [-0.55 to 0.03], Standard Error of Mean 0.14

6. Secondary Outcome: Duration of Hospitalization/Per Patient
Description: Over the 12 months of the study we calculated mean duration of hospitalization/per patients.
Time Frame: 12 months
Measure: Mean (Standard Error); unit: day/per patient
Arm/Group | Broncho-Vaxom Group | Placebo Group
Number analyzed (Participants) | 35 | 40
day/per patient | 0.82 (0.35) | 2.02 (0.71)
Statistical Analysis 1: Comparison: Broncho-Vaxom Group vs Placebo Group; Test type: Superiority or Other; p = 0.452, Wilcoxon (Mann-Whitney) — P value was not need to adjusted for multiple comparisons; Mean Difference (Final Values) = -1.22, 95% CI 2-sided [-2.87 to 0.42], Standard Error of Mean 0.82

7. Secondary Outcome: Effect of OM-85 BV on Cytokine Levels
Description: Cytokine levels were not measured during the trial because of unavailability of laboratory resources.
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Description: 3 patients receiving OM-85, and 2 patients receiving placebo reported 5 adverse reactions.These were diarrhea (1 patient), abdominal pain (1 patient) and erythema nodosum (one patient) in the OM-85 group and diarrhea (1 patient), abdominal pain (1 patient) in the placebo group.
Arm/Group | Broncho-Vaxom Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/40
Other Adverse Events (participants affected / at risk) | 3/35 | 2/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Broncho-Vaxom Group (N=35) | Placebo Group (N=40)
diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
erythema nodosum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Main shortcoming of our study is the small sample size. This might have hampered the appearance of some statistically meaningful differences such as wheezing attacks that require steroid treatment, rate and duration of hospitalizations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No